CLINICAL TRIAL: NCT00028678
Title: A Phase II Study to Evaluate the Effect of Dalteparin and Radiation Therapy on Survival Compared to the RTOG RPA Database and on Thromboembolic Events in Patients With Newly Diagnosed Glioblastoma Multiforme
Brief Title: Dalteparin and Radiation Therapy in Treating Patients With Newly Diagnosed Supratentorial Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Group Chair, Eastern Cooperative Oncology Group
Purpose: Treatment
Other Study IDs: CDR0000069119; E1F01
Record Dates: First submitted 2002-01-04; First posted 2003-02-06 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Dalteparin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: dalteparin
Radiation: radiation therapy

SUMMARY:
RATIONALE: Dalteparin may stop the growth of cancer by stopping blood flow to the tumor and by blocking the enzymes necessary for tumor cell growth. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining dalteparin with radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining dalteparin with radiation therapy in treating patients who have newly diagnosed supratentorial glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether dalteparin, initiated at the time of conventional radiotherapy, improves the median survival of patients with newly diagnosed supratentorial glioblastoma multiforme.
* Determine the time to progression in patients treated with this regimen.
* Determine the incidence of thromboembolic events in patients treated with this regimen.
* Determine the feasibility and toxicity of dalteparin in this patient population.

OUTLINE: This is a multicenter study.

Patients undergo cranial irradiation 5 days a week for 7 weeks. Beginning concurrently with initiation of radiotherapy, patients receive dalteparin subcutaneously once daily for up to 2 years in the absence of unacceptable toxicity. Patients may continue receiving dalteparin after year 2 at the discretion of the investigator.

Patients are followed every 3 months for 2 years and then every 6 months for up to 5 years after study entry.

PROJECTED ACCRUAL: A total of 72 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed newly diagnosed supratentorial glioblastoma multiforme
* At least 2 weeks but no more than 4 weeks since prior surgery

  * Patients with biopsy only must be at least 1 week past surgery

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Platelet count at least 100,000/mm^3
* No history of heparin-induced thrombocytopenia
* No coagulopathy

Hepatic:

* Bilirubin no greater than 2.5 mg/dL
* AST no greater than 3 times upper limit of normal (ULN)
* PT/aPTT no greater than 1.5 times ULN

Renal:

* Creatinine no greater than 2.0 mg/dL
* No gross hematuria within the past 6 months

Cardiovascular:

* No uncontrolled hypertension
* No unstable angina
* No symptomatic congestive heart failure
* No myocardial infarction within the past 6 months
* No uncontrolled cardiac arrhythmia

Gastrointestinal:

* No peptic ulcer disease within the past 6 months
* Negative stool guaiac

  * Negative endoscopy required if positive stool guaiac

Other:

* No known hypersensitivity to dalteparin, heparin, or pork products
* No CNS trauma within the past 3 months
* No intracranial or intraocular hemorrhage, unless related to surgery, within the past 6 months
* No retinal detachment within the past 6 months
* No other concurrent malignancy receiving treatment
* No active infection
* No AIDS-related illness
* HIV negative
* Must weigh at least 90 pounds (40 kg)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunomodulators
* No concurrent investigational matrix metalloproteinase inhibitors or antiangiogenesis agents

Chemotherapy:

* Prior chemotherapy for other malignancy allowed
* No concurrent standard or investigational cytotoxic chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior cranial irradiation
* Prior radiotherapy for other malignancy allowed
* Concurrent radiotherapy allowed

Surgery:

* See Disease Characteristics
* Recovered from prior surgery
* No prior eye or ear surgery

Other:

* No concurrent nonsteroidal anti-inflammatory drugs
* No ongoing or concurrent aspirin or anticoagulation therapy except routine central venous catheter flushing
* No other concurrent non-protocol therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2002-07-11 (Actual); Primary Completion 2006-07 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. I. Robins, MD, PhD, Study Chair — University of Wisconsin, Madison
Locations (12):
- United States (12):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - CCOP - Scott and White Hospital, Temple, Texas
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- [Result] Robins HI, O'Neill A, Gilbert M, Olsen M, Sapiente R, Berkey B, Mehta M. Effect of dalteparin and radiation on survival and thromboembolic events in glioblastoma multiforme: a phase II ECOG trial. Cancer Chemother Pharmacol. 2008 Jul;62(2):227-33. doi: 10.1007/s00280-007-0596-3. Epub 2007 Sep 20. PMID 17882417